CLINICAL TRIAL: NCT02713594
Title: Wisconsin Tobacco Quit Line Centers for Medicaid Services Striving To Quit Evaluation Project
Brief Title: Wisconsin Tobacco Quit Line Medicaid Incentive Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-0056 (400025710)
Record Dates: First submitted 2016-02-16; First posted 2016-03-18 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Smoking; Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Counseling from WTQL
  Interventions: Behavioral: Counseling from WTQL
- Incentive (Experimental): Counseling from WTQL; Financial incentive to participate
  Interventions: Behavioral: Counseling from WTQL; Other: Financial incentive to participate

INTERVENTIONS:
Behavioral: Counseling from WTQL — Counseling from the Wisconsin Tobacco Quit Line (WTQL) consisted of 5 proactive calls to the participant to help them successfully quit tobacco use, plus ad hoc calls at the participant's initiation; also, WTQL coaches encouraged participants to see their health care provider to obtain Medicaid-approved smoking cessation medications to help them quit smoking.
Other: Financial incentive to participate — Participants in the Incentive condition received $30 per call for up to five WTQL calls taken; in addition, Incentive condition participants received $40 for producing biochemical evidence of abstinence at the 6-month follow-up visit. (Note that participants in both the Control condition and the Incentive condition received $40 for completing the baseline biochemical smoking status assessment visit and $40 for completing the 6-month follow-up biochemical smoking status assessment visit.) Compensation was in the form of prepaid Visa gift cards mailed approximately 2-4 weeks after the point of contact.
  Arms: Incentive

SUMMARY:
The study is designed to test the hypotheses that financial incentives can increase both participation in smoking cessation treatment and resulting cessation rates, when they are offered to BadgerCare Plus (Medicaid) smokers as part of their health care.

DETAILED DESCRIPTION:
Previous research on providing incentives for healthy behaviors has shown that financial incentives can increase treatment participation and boost outcomes when they are tied to participation in evidence based treatments. However, most of this research has been done in laboratory settings and in relatively small clinical trials. This study is designed to test the hypotheses that incentives can increase both participation in smoking cessation treatment and resulting cessation rates, when they are offered to Wisconsin BadgerCare Plus (Medicaid) smokers as part of their health care. If successful, this treatment approach could be used more broadly to reduce the considerable financial and personal costs associated with smoking-related disease.

In this study, Medicaid-eligible smokers were recruited from primary care clinics and from callers to the Wisconsin Tobacco Quit Line (WTQL) with randomization a Control condition and an Incentive condition. All participants were offered five cessation calls from the WTQL and participants were encouraged by WTQL coaches to obtain cessation medication from their primary care providers. All participants received payment for completing a baseline assessment ($40) and a 6-month smoking test ($40). Only Incentive condition participants received additional compensation for taking counseling calls ($30 per completed call) and for biochemically-verified abstinence at the 6-month visit ($40).

ELIGIBILITY:
Inclusion Criteria:

* enrollment in Wisconsin Medicaid (BadgerCare Plus)
* resides in study area (one of 25 counties)
* 18 or older
* English or Spanish speaking
* has smoked daily (at least 5 cigarettes each day) over the last week
* willingness to attend visits at his/her PCC (primary care clinic) or go to a testing site at baseline and 6 months (2 times over a 6 month period), provide urine samples or participate in exhaled carbon monoxide testing, and complete follow-up phone calls from the WTQL
* willingness to inform the WTQL as to any change in address, phone number, clinic attended, or health plan.

Exclusion Criteria:

* not enrolled in Wisconsin Medicaid (BadgerCare Plus)
* not reside in study area
* less than 18 years of age
* not English or Spanish speaking
* does not smoke daily (at least 5 cigarettes each day) over the last week
* not willing to attend visits at his/her PCC (primary care clinic) or alternative testing site at baseline and 6 months (2 times over a 6 month period), provide urine or exhaled carbon monoxide samples, and complete follow-up phone calls.
* not willing to inform the WTQL as to any change in address, phone number, clinic attended, or health plan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy b Baker, PhD, Principal Investigator — University of Wisconsin--CTRI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraser DL, Fiore MC, Kobinsky K, Adsit R, Smith SS, Johnson ML, Baker TB. A Randomized Trial of Incentives for Smoking Treatment in Medicaid Members. Am J Prev Med. 2017 Dec;53(6):754-763. doi: 10.1016/j.amepre.2017.08.027. Epub 2017 Nov 2. PMID 29079405

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants in the Control condition received counseling from the Wisconsin Tobacco Quit Line (WTQL) consisting of 5 proactive calls to the participant to help them successfully quit tobacco use, plus ad hoc calls at the participant's initiation; also, WTQL coaches encouraged participants to see their health care provider to obtain Medicaid-approved smoking cessation medications to help them quit smoking.
- Incentive: Participants in the Incentive Condition received counseling from the Wisconsin Tobacco Quit Line (WTQL) consisting of 5 proactive calls to the participant to help them successfully quit tobacco use, plus ad hoc calls at the participant's initiation; also, WTQL coaches encouraged participants to see their health care provider to obtain Medicaid-approved smoking cessation medications to help them quit smoking.
  Participants in the Incentive condition also received financial incentives to complete proactive counseling calls from the WTQL received ($30 per completed call); in addition, Incentive condition participants received $40 for producing biochemical evidence of abstinence at the 6-month follow-up visit.
Period: Overall Study
Arm/Group | Control | Incentive
Started | 952 | 948
Completed | 562 | 552
Not Completed | 390 | 396
Not completed — Withdrawal by Subject | 32 | 22
Not completed — Lost to Follow-up | 358 | 374

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Incentive | Total
Number analyzed (Participants) | 952 | 948 | 1900
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.2) | 45.0 (11.2) | 45.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 577 | 569 | 1146
  Male | 375 | 379 | 754
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 390 | 393 | 783
  Black or African American | 487 | 485 | 972
  Asian | 3 | 1 | 4
  American Indian/Alaska Native | 18 | 16 | 34
  Other | 36 | 38 | 74
  Refused/Do not know/Not collected | 18 | 15 | 33
Region of Enrollment [Number; unit: Count of Participants]
  United States | 952 | 948 | 1900

OUTCOME MEASURES:

1. Primary Outcome: Abstinence From Smoking
Description: The primary outcome data will be the biochemically confirmed abstinence using urine (measured cotinine) or exhaled (breath) carbon monoxide (CO).
Time Frame: Measured 6 months after enrollment at follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Incentive
Number analyzed (Participants) | 952 | 948
Participants | 131 | 205
Statistical Analysis 1: Comparison: Control vs Incentive; Test type: Superiority or Other; p < .0001, Abstinence Risk Difference; Risk Difference (RD) = -7.86, 95% CI 2-sided [-11.28 to -4.5]

2. Secondary Outcome: Engagement in Treatment
Description: This analysis will compare number of calls completed
Time Frame: Measured 6 months after enrollment at follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Incentive
Number analyzed (Participants) | 952 | 948
Participants
  Zero Calls Taken | 6 | 3
  1 Call Taken | 245 | 76
  2 Calls Taken | 179 | 113
  3 Calls Taken | 154 | 122
  4 Calls Taken | 165 | 199
  5 Calls Taken | 203 | 435
Statistical Analysis 1: Comparison: Control vs Incentive; Test type: Superiority or Other; p < .0001, Chi-squared; Chi-square test value = 196.1, with 5 degrees of freedom

3. Secondary Outcome: Cost-effectiveness
Description: This analysis will quantify the costs of treatment for Control and Incentive conditions with regard to attaining 6-month abstinence. Project costs were allocated to three categories: 1) Service costs, including billed staff time for counseling and testing, as well as all incidentals connected with services; 2) Incentives and distribution costs; and 3) Service-related administrative costs, including promotion/marketing and staff time for administering the intervention. Costs of planning the project, grant administration, and research within the project are not included in the analysis.The outcome is the cost per quit in each treatment group. Cost per quit in each group was calculated by: 1) computing the grand total of costs for all participants in a given group; and 2) dividing the grand total for a given group by the number of successful quitters. As such, the cost per quit is a single value with no measure of dispersion.
Time Frame: Measured 6 months after enrollment
Measure: Number; unit: U.S. Dollars
Groups:
- Incentive: Counseling from WTQL; Financial incentive to participate
  Counseling from WTQL: Counseling from the Wisconsin Tobacco Quit Line (WTQL) consisted of 5 proactive calls to the participant to help them successfully quit tobacco use, plus ad hoc calls at the participant's initiation; also, WTQL coaches encouraged participants to see their health care provider to obtain Medicaid-approved smoking cessation medications to help them quit smoking.
  Financial incentive to participate: Participants in the Incentive condition received $30 per call for up to five WTQL calls taken; in addition, Incentive condition participants received $40 for producing biochemical evidence of abstinence at the 6-month follow-up visit. (Note that participants in both the Control condition and the Incentive condition received $40 for completing the baseline biochemical smoking status assessment visit and $40 for completing the 6-month follow-up biochemical smoking status assessment visit.)
Arm/Group | Control | Incentive
Number analyzed (Participants) | 952 | 948
U.S. Dollars | 5193 | 4108

ADVERSE EVENTS:
Description: Adverse event data were not collected as per study protocol; no study medications were part of the protocol.
Arm/Group | Control | Incentive
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No